CLINICAL TRIAL: NCT02272140
Title: A Prospective, Non-randomized, Multicenter Evaluation of the Utility of Transcutaneous Stimulation of the Lumbosacral Nerve Roots During XLIF® and Its Relationship to Postoperative Nerve Health
Brief Title: Advanced XLIF Monitoring Multicenter Study
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.NV1401
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Lumbar Disc Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the utility of localized stimulation of the lumbosacral nerve roots during XLIF through correlation of observed changes in the response latency, amplitude, waveform morphology, and/or response threshold with surgical events. Additionally, correlation between neuromonitoring findings and postoperative neural status will be evaluated.

DETAILED DESCRIPTION:
The utility of NVM5 neuromonitoring by stimulating within the surgical site during XLIF has been previously demonstrated; however, it is possible that depending on the site of injury, this method of monitoring may stimulate nerves at a location that is distal to the site of injury along the nerve conduction pathway. In this example, the site of injury would not disrupt the stimulus and a normal muscle response may occur, providing a false negative result. With this in mind, it has been hypothesized that more accurate information may be gathered by stimulating the lumbar roots or spinal nerves cranial to the surgical site and recording the subsequent muscle response in the lower limbs. Using this technique, the response to the stimulus would traverse the surgical site, including the site of any nerve injury. Currently, the only described method of stimulating cranial to the surgical site is with transcranial motor evoked potentials (tcMEP); stimulating the lumbosacral nerve roots locally has not been demonstrated. Though tcMEP monitoring is a well-documented technique, there are several limitations associated with its use. For example, tcMEP requires adherence to total intravenous anesthesia (TIVA), thereby restricting the use of inhalational agents. This restriction may require additional training and coordination with the anesthesiologist, as well as added cost to the hospital.6 Additional challenges with tcMEP include the requirements for high voltage stimulation to successfully transmit a stimulus across the skull. In rare instances this can cause seizures, tongue lacerations, and other complications. Finally, due to inclusion of the central nervous system, monitoring with tcMEP may be less reproducible and specific than a more localized stimulation.

To address these challenges, recent adaptations to standard MEP and EMG monitoring protocols have used local stimulation of the lumbosacral nerve roots at the level of the conus, with recorded responses from the relevant innervated muscle groups of the lower limbs. Early experience using this technique has shown the feasibility and reproducibility of obtaining reliable baseline and longitudinal responses throughout a surgical procedure, and incorporation of this monitoring modality has become common practice at certain surgical sites performing XLIF, although determination of clinically meaningful changes in those responses have yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female spine surgery patients who are at least 18 years of age;
2. Persistent back and/or leg pain unresponsive to conservative treatment for at least six (6) months, unless surgical treatment is clinically indicated earlier;
3. Surgical candidates for extreme lateral approach lumbar spine surgery at spinal levels L2 to L5, inclusive of L4-5;
4. Able to undergo surgery based on physical exam, medical history and surgeon judgment;
5. Patients who understand the conditions of enrollment and are willing to sign an informed consent to participate in the evaluation.

Exclusion Criteria:

1. Patient has a mental or physical condition that would limit the ability to comply with study requirements;
2. Currently undergoing any surgical treatment at any spinal level other than L2 to L5;
3. Currently undergoing surgical treatment for significant deformity correction (e.g., osteotomy, anterior longitudinal ligament release, or other significant manipulation of the spinal column);
4. Underlying neurological disease or neurological deficit that is not associated with the condition for which he/she is seeking surgical intervention (e.g., diabetic peripheral neuropathy);
5. Implanted pacemaker, defibrillator, or other electronic devices;
6. Involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested);
7. Pregnant women;
8. Patient is a prisoner;
9. Patient is participating in another clinical study that would confound study data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who, in the investigator's opinion, require lateral approach spinal fusion surgery at spinal level L4-5 (though may include any number of levels from L2 through L5), and have consented to XLIF surgery for their condition will be included. All subjects must meet the inclusion/exclusion criteria below in order to be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of this neuromonitoring technique in identifying neural injury after the XLIF procedure. | 6 weeks
  Intraoperative neuromonitoring findings will be correlated with postoperative neural status up to six weeks post-op to determine the sensitivity and specificity of this testing modality's ability to detect postoperative decreases in motor function during the XLIF procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — NuVasive
Locations (12):
- United States (12):
  - Scripps Clinical Research Services, La Jolla, California
  - USF Neurology and Neurosurgery, Tampa, Florida
  - Foundation for Orthopaedic Research and Education (FORE), Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - West Augusta Spine Specialists, LLC, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia Orthopedic Group Research, Columbia, Missouri
  - Western Regional Center for Brain & Spine Surgery, Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seton Brain and Spine Institute, Austin, Texas
  - Northwest Orthopaedic Specialists, P.S., Spokane, Washington

IPD SHARING:
Plan to Share IPD: No